CLINICAL TRIAL: NCT01444924
Title: Transversus Abdominis Plane Blocks for Patients Undergoing Robotic Gynecologic Oncology Surgery: A Prospective Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Transversus Abdominis Plane Blocks for Patients Undergoing Robotic Gynecologic Oncology Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2011-0274; CO11701 (Other: UWCCC); 2011-0274 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH\OBSTET & GYNECOL ONC (Other: UW Madison); NCI-2011-03675 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2018-03

CONDITIONS: Gynecologic Cancer; Post-operative Pain
Keywords: Pain control; Gynecologic Oncology; Surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivicaine (Experimental): TAP block with bupivicaine/epinephrine placed prior to surgery.
  Interventions: Drug: Bupivicaine
- Placebo (Placebo Comparator): TAP block with placebo placed prior to surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivicaine — The TAP block will be placed using a standardized ultrasound-guided approach. Subjects assigned to the study group will have an injection of 30 mL 0.25% bupivacaine, a local anesthetic with 3 mcg/mL of epinephrine, placed into the plane between the internal oblique and the transversus abdominis
  Arms: Bupivicaine
Drug: Placebo — The placebo block will be placed in a similar manner, using a standardized ultrasound-guided approach. The placebo injection will consist of 30 mL sterile, preservative-free saline.
  Arms: Placebo

SUMMARY:
This study is a single-center, randomized, placebo-controlled, double-blind clinical trial. The purpose of this study is to evaluate the impact of pre-operative transverses abdominis plane (TAP) blocks on post-operative analgesia in patients undergoing robotic surgery for gynecologic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robotic-assisted surgery under the care of the Division of Gynecologic Oncology at UWHC.
* Patients must be ≥18 years old.
* Patients must be English speaking.
* Patients must have the ability to understand visual and verbal pain scales.
* ASA physical status 1-3.

Exclusion Criteria:

* Known allergy to local anesthetics.
* Immunocompromised.
* Known history of opioid dependence, as available within the medical record and standard of care pre-operative work-up.
* Known history of chronic pain disorders.
* Pregnancy or lactation.
* Patient is a prisoner or incarcerated.
* Significant liver disease that would inhibit prescription of opioids.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 75 patients agreed to participate in the study. Eight patients did not meet inclusion criteria for the study, 2 patients were excluded from the analysis secondary to intraoperative conversion to laparotomy, and 1 additional patient was excluded because the robot was unavailable. This left a total of 64 subjects who completed the study.
Period: Overall Study
Arm/Group | Bupivicaine | Placebo
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treatment group, who received TAP block placement, was younger than the saline injection group, on average (55.2 versus 62.1, P = 0.028).
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivicaine | Placebo | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.48) | 62.1 (14.29) | 58.7 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 31 | 29 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.2 (12.12) | 36.3 (9.01) | 35.3 (12.32)

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Post Operative Opioid Consumption, Converted to Intravenous Morphine Equivalents
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Bupivicaine | Placebo
Number analyzed (Participants) | 31 | 33
mg | 64.9 (28.65) | 69.3 (32.73)

2. Secondary Outcome: Pain Scores
Description: Pain scores by the Visual Analog Scale (VAS) [0-5, where 0 is no pain and 5 is extreme] and Wisconsin Brief Pain Inventory (BPI) [where 0 is no pain and 10 is the most painful], will be collected 3 times post-operatively (once the day of surgery (at least 2 hours post-op) and both the morning and afternoon/evening on post-operative day #1). Pain scores will be analyzed individually using the chi-squared test and linear regression. All statistical calculations used a two-sided significance level of 0.05 and were calculated using the R Project for Statistical Computing. VAS and BPI scores for each subject were averaged to provide a resultant VAS and BPI score.
Time Frame: from 2 hours post-op to the afternoon/evening of post-op day #1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bupivicaine | Placebo
Number analyzed (Participants) | 31 | 33
units on a scale
  VAS | 3.12 [2.48 to 3.76] | 3.61 [2.88 to 4.35]
  BPI | 6.44 [5.56 to 7.32] | 6.97 [6.15 to 7.79]

ADVERSE EVENTS:
Time Frame: 2-4 weeks post-op
Arm/Group | Bupivicaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

LIMITATIONS AND CAVEATS:
Unilateral placement of block may decrease overall effectiveness. Sample size was small, from single institution, and encompassed a variety of diagnoses and procedures. Analysis also included intraoperative medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No